CLINICAL TRIAL: NCT00168779
Title: A Randomized, Double-blind, Placebo-controlled, Forced-titration, Phase IV Study Comparing Telmisartan 80 mg + Hydrochlorothiazide 25 mg Versus Valsartan 160 mg + Hydrochlorothiazide 25 mg Taken Orally for Eight Weeks in Patients With Stage 1 or Stage 2 Hypertension.
Brief Title: Randomized, Double-Blind, Placebo-Controlled, Forced-Titration, Comparing Telmisartan vs Valsartan. Taken Orally for Eight Weeks in Patients With Stage 1 and Stage 2 Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 502.476
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide; Valsartan

INTERVENTIONS:
Drug: telmisartan 80 mg / hydrochlorothiazide 25 mg
Drug: valsartan 160 mg / hydrochlorothiazide 25 mg
Drug: placebo

SUMMARY:
The primary objective of this study is to compare the effectiveness of telmisartan 80 mg / hydrochlorothiazide 25 mg [Micardis HCT] to valsartan 160 mg / hydrochlorothiazide 25 mg [Diovan HCT] and placebo in the treatment of Stage 1 and Stage 2 hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Age 18 years or older
3. Ability to stop current antihypertensive therapy without unacceptable risk to the patient (investigator's discretion)
4. Seated cuff DBP of ? 95 mmHg at Visit 2 (baseline)

Exclusion Criteria:

1. Pre-menopausal women (last menstruation ? 1 year prior to start of run-in period) who:

   1. are not surgically sterile and/or
   2. are nursing or pregnant
   3. are of child-bearing potential and are NOT practicing acceptable means of birth control, do NOT plan to continue using this method throughout the study and do NOT agree to submit to periodic pregnancy testing during participation in studies of > 3-months duration. Acceptable methods of birth control include oral, implantable, transdermal, or injectable contraceptives, and Intra-Uterine Device (IUD).
2. Known or suspected secondary hypertension.
3. Mean seated SBP >= 180 mmHg or mean seated DBP >= 120 mmHg during any clinic visit prior to randomization.
4. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   1. SGPT (ALT) or SGOT (AST) > 2 times the upper limit of normal range, or
   2. Serum creatinine > 3.0 mg/dL or creatinine clearance < 0.6 ml/sec.
5. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant or with only one kidney.
6. Clinically relevant hypokalemia or hyperkalemia.
7. Uncorrected volume depletion.
8. Uncorrected sodium depletion.
9. Primary aldosteronism.
10. Hereditary fructose intolerance.
11. Biliary obstructive disorders, cholestatis or moderate to severe hepatic in sufficiency.
12. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists.
13. History of drug or alcohol dependency within six months prior to start of run-in period.
14. Chronic administration of any medications known to affect blood pressure, exc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1185
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Mean seated trough cuff DBP and SBP | after 8 week

SECONDARY OUTCOMES:
The percentage of patients responding to treatment based on in-clinic mean seated trough cuff measurements | after 8 week
The percentage of patients with uncontrolled hypertension | after 8 weeks
Change in the in-clinic mean seated cuff DBP and SBP at the one and three hour post dose time points | after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (113):
- United States (113):
  - 502.476.074 Boehringer Ingelheim Investigational Site, Athens, Alabama
  - 502.476.059 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 502.476.071 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 502.476.079 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 502.476.014 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 502.476.031 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 502.476.110 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 502.476.037 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 502.476.061 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 502.476.066 Boehringer Ingelheim Investigational Site, Carlisle, Arkansas
  - 502.476.067 Boehringer Ingelheim Investigational Site, Buena Park, California
  - 502.476.086 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 502.476.124 Boehringer Ingelheim Investigational Site, Greenbrae, California
  - 502.476.005 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 502.476.024 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 502.476.029 Boehringer Ingelheim Investigational Site, Redondo Beach, California
  - 502.476.048 Boehringer Ingelheim Investigational Site, Riverside, California
  - 502.476.073 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 502.476.087 Boehringer Ingelheim Investigational Site, San Diego, California
  - 502.476.111 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 502.476.050 Boehringer Ingelheim Investigational Site, Santa Ana, California
  - 502.476.026 Boehringer Ingelheim Investigational Site, Spring Valley, California
  - 502.476.033 Boehringer Ingelheim Investigational Site, Tulsa, California
  - 502.476.019 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 502.476.101 Boehringer Ingelheim Investigational Site, Highlands Ranch, Colorado
  - 502.476.053 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 502.476.032 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 502.476.041 Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - 502.476.108 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 502.476.015 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 502.476.044 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 502.476.058 FPA Clinical Research, Kissimmee, Florida
  - 502.476.052 Boehringer Ingelheim Investigational Site, Largo, Florida
  - 502.476.080 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 502.476.021 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 502.476.012 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 502.476.036 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 502.476.065 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 502.476.022 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 502.476.049 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 502.476.008 Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - 502.476.075 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 502.476.018 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 502.476.047 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 502.476.004 Boehringer Ingelheim Investigational Site, Peoria, Illinois
  - 502.476.062 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 502.476.063 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 502.476.051 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 502.476.084 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 502.476.090 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 502.476.100 Boehringer Ingelheim Investigational Site, Newton, Kansas
  - 502.476.003 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 502.476.038 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 502.476.002 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 502.476.116 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 502.476.035 Boehringer Ingelheim Investigational Site, Oxon Hill, Maryland
  - 502.476.010 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 502.476.028 Boehringer Ingelheim Investigational Site, Brooklyn Center, Minnesota
  - 502.476.057 Boehringer Ingelheim Investigational Site, Edina, Minnesota
  - 502.476.055 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 502.476.114 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 502.476.112 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 502.476.126 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 502.476.125 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 502.476.120 Boehringer Ingelheim Investigational Site, Berlin, New Jersey
  - 502.476.088 Boehringer Ingelheim Investigational Site, Ship Bottom, New Jersey
  - 502.476.089 Boehringer Ingelheim Investigational Site, Turnersville, New Jersey
  - 502.476.068 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 502.476.122 Boehringer Ingelheim Investigational Site, Hamburg, New York
  - 502.476.020 Boehringer Ingelheim Investigational Site, Northport, New York
  - 502.476.025 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 502.476.091 Boehringer Ingelheim Investigational Site, Williamsville, New York
  - 502.476.046 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 502.476.083 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 502.476.042 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 502.476.095 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 502.476.027 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 502.476.034 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 502.476.060 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 502.476.016 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 502.476.023 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 502.476.128 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 502.476.064 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 502.476.103 Boehringer Ingelheim Investigational Site, Olmsted Falls, Ohio
  - 502.476.007 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 502.476.113 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 502.476.030 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 502.476.104 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 502.476.109 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 502.476.094 Boehringer Ingelheim Investigational Site, Harleysville, Pennsylvania
  - 502.476.121 Boehringer Ingelheim Investigational Site, Penndel, Pennsylvania
  - 502.476.072 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 502.476.076 Boehringer Ingelheim Investigational Site, Springfield, Pennsylvania
  - 502.476.013 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 502.476.085 Boehringer Ingelheim Investigational Site, Cordova, Tennessee
  - 502.476.096 Boehringer Ingelheim Investigational Site, Jackson, Tennessee
  - 502.476.081 Boehringer Ingelheim Investigational Site, New Tazewell, Tennessee
  - 502.476.082 Boehringer Ingelheim Investigational Site, Selmer, Tennessee
  - 502.476.039 Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - 502.476.056 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 502.476.069 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 502.476.107 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 502.476.070 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 502.476.001 Boehringer Ingelheim Investigational Site, Bountiful, Utah
  - 502.476.006 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 502.476.017 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 502.476.097 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 502.476.098 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 502.476.011 Boehringer Ingelheim Investigational Site, Falls Church, Virginia
  - 502.476.093 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 502.476.078 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 502.476.106 Boehringer Ingelheim Investigational Site, Menomonee Falls, Wisconsin
  - 502.476.105 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/22844584